CLINICAL TRIAL: NCT05309551
Title: The Effects of Inspiratory Muscle Training Immediatley After Lung Transplantation: a Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training Immediately After Lung Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Cristiane Meirelles, PT, PhD, Associate Professor-Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021H0310
Record Dates: First submitted 2022-03-22; First posted 2022-04-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lung Transplantation; Chronic Lung Disease; Muscle Weakness; Rehabilitation
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Inspiratory Muscle training- Intervention group (Experimental): Along with standard post-transplant physical therapy, the intervention group will begin daily respiratory exercise training utilizing the IMT trainer device (POWERbreathe Medic Plus®) with weekly incremental increases in respiratory load. Patients will be asked to use the IMT device twice per day, 7 days per week, for 8 weeks.
  Interventions: Device: IMT- Intervention group
- Inspiratory Muscle training - Placebo group (Sham Comparator): Along with standard post-transplant physical therapy, the placebo group will begin daily respiratory exercise training utilizing the IMT trainer device (POWERbreathe Medic Plus®) with no increase of respiratory load. Patients will be asked to use the IMT device twice per day, 7 days per week, for 8 weeks.
  Interventions: Device: IMT- Placebo group
- Usual care group (No Intervention): Patients will only participate in standard post-transplant physical therapy.

INTERVENTIONS:
Device: IMT- Intervention group — The resistive load will be readjusted weekly to reach 50% of maximal inspiratory pressure (MIP).
  Other Names: POWERBreathe Medic Plus®
  Arms: Inspiratory Muscle training- Intervention group
Device: IMT- Placebo group — The inspiratory resistive load will be adjusted to the minimum value of the device (9 cm H2O) during all inspiratory muscle training sessions.
  Other Names: POWERBreathe Medic Plus®
  Arms: Inspiratory Muscle training - Placebo group

SUMMARY:
Following lung transplantation (LTX), patients may exhibit respiratory and skeletal muscle weakness that will affect exercise capacity, increase dyspnea and fatigue, limit activities of daily living (ADL) and decrease quality of life.

Inspiratory muscle training (IMT) has been extensively studied in a variety of non-LTX populations and research has shown that IMT improves exercise capacity, diaphragmatic thickness, and reduced dyspnea during activities of daily living and improved quality of life in patients with advanced lung disease.

The aim of this randomized controlled study is to investigate the benefits of providing inspiratory muscle training via use of an inspiratory muscle trainer device in addition to standard physical therapy in the acute phase of rehabilitation following LTX. Patients targeted for enrollment will be those with any type of advanced lung disease requiring LTX with the objective of demonstrating improvements in respiratory muscle recovery, perceived dyspnea, severity of fatigue, and overall functional status following the transplant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant has personally signed and dated informed consent form indicating understanding of all pertinent aspects of the study
* Active on the waiting list for lung transplantation
* Able to ambulate pre-transplant (not bed/wheelchair bound) with or without assistive device

Exclusion Criteria:

* Already participating in a regular IMT program
* Impaired cognition with inability to follow commands

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in inspiratory muscle strength: Maximal inspiratory pressure (MIP) measured in cmH2O | The groups will be assessed: Before Lung transplantation, at baseline (immediate post-transplant), 8 weeks, 6 and 12 months after LTX
  Inspiratory muscle strength will be measured as maximal inspiratory pressure (MIP) using a POWERbreathe® KH2, International Ltd; UK. The MIP is defined as the greatest negative pressure sustained for at least one second by each patient. The patient will be verbally encouraged to perform three to five inspiratory maneuvers at maximal intensity. The maximum value will be used for the analysis.
Change in perceived dyspnea: Modified Medical Research Council Dyspnea Scale | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Modified Medical Research Council Dyspnea Scale (mMRC) will measure dyspnea perceptions during the activities of daily living. A score from 0-4 is used to classify the impact of dyspnea on physical function in patients with respiratory limitations. 0 represents a person who suffers from dyspnea only with strenuous exercise. 4 represents a person who are too breathless to leave the house, or breathless when dressing.
Change in fatigue: Fatigue Severity Scale | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Fatigue Severity Scale (FSS) evaluates fatigue using a nine-item, self-scored questionnaire, which with a visual ranking format ranging from one to seven that quantifies patient-perceived fatigue. Higher composite scores indicate more severe fatigue. An average score of less than 2.8 indicates no fatigue, and more than 6.1 indicates chronic fatigue syndrome.
Change in functional capacity | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Functional capacity will be estimated using the 6-minute walk test according to the American Thoracic Society guidelines. Before and after the test, oxygen saturation (SpO2), heart rate, Modified Dyspnea Borg Scale and walking distance will be recorded

SECONDARY OUTCOMES:
Change in lung function: Pulmonary Function Test | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Lung function will be measured in accordance with the guidelines of the American Thoracic Society. The following variables will be analyzed: (a) forced vital capacity (FVC, L) and (b) forced expiratory volume in the first second (FEV1, L).
Change in physical performance | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Physical performance test will be evaluated using the Short Physical Performance Battery Test (SPPB) to assess standing balance, walking speed, and chair stands. The corresponding score from each section is determined and compiled for an overall score of 0-12.
Change in lower extremity muscle strength | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Quadriceps strength will be measured with a hand-held dynamometer (HHD, Microfet®, Hogan Health Industries, Inc., UT, USA). At least three measurements will be obtained and the higher knee extensor muscle strength value will be used for the analysis.
Change in grip strength | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Grip strength will be performed using a digital dynamometer. At least three measurements will be obtained and the highest reproducible value will be taken into analysis and related to reference values.
Change in quality of life | The groups will be assessed: Before Lung transplantation, 8 weeks, 6 and 12 months after LTX
  Heath related quality of life will be measured using the SF-36 questionnaire. The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH).

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Meirelles, PT, PhD, Principal Investigator — School of Health and Rehabilitation Sciences- Physical Therapy Division
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brocki BC, Andreasen JJ, Langer D, Souza DS, Westerdahl E. Postoperative inspiratory muscle training in addition to breathing exercises and early mobilization improves oxygenation in high-risk patients after lung cancer surgery: a randomized controlled trial. Eur J Cardiothorac Surg. 2016 May;49(5):1483-91. doi: 10.1093/ejcts/ezv359. Epub 2015 Oct 20. PMID 26489835
- [Background] Hanada M, Kasawara KT, Mathur S, Rozenberg D, Kozu R, Hassan SA, Reid WD. Aerobic and breathing exercises improve dyspnea, exercise capacity and quality of life in idiopathic pulmonary fibrosis patients: systematic review and meta-analysis. J Thorac Dis. 2020 Mar;12(3):1041-1055. doi: 10.21037/jtd.2019.12.27. PMID 32274173
- [Background] Bissett B, Gosselink R, van Haren FMP. Respiratory Muscle Rehabilitation in Patients with Prolonged Mechanical Ventilation: A Targeted Approach. Crit Care. 2020 Mar 24;24(1):103. doi: 10.1186/s13054-020-2783-0. PMID 32204719
- [Background] Hoffman M, Augusto VM, Eduardo DS, Silveira BMF, Lemos MD, Parreira VF. Inspiratory muscle training reduces dyspnea during activities of daily living and improves inspiratory muscle function and quality of life in patients with advanced lung disease. Physiother Theory Pract. 2021 Aug;37(8):895-905. doi: 10.1080/09593985.2019.1656314. Epub 2019 Aug 20. PMID 31429627
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Evans JA, Whitelaw WA. The assessment of maximal respiratory mouth pressures in adults. Respir Care. 2009 Oct;54(10):1348-59. PMID 19796415
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bernabeu-Mora R, Medina-Mirapeix F, Llamazares-Herran E, Garcia-Guillamon G, Gimenez-Gimenez LM, Sanchez-Nieto JM. The Short Physical Performance Battery is a discriminative tool for identifying patients with COPD at risk of disability. Int J Chron Obstruct Pulmon Dis. 2015 Dec 3;10:2619-26. doi: 10.2147/COPD.S94377. eCollection 2015. PMID 26664110
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Talwar A, Sahni S, John S, Verma S, Cardenas-Garcia J, Kohn N. Effects of pulmonary rehabilitation on Fatigue Severity Scale in patients with lung disease. Pneumonol Alergol Pol. 2014;82(6):534-40. doi: 10.5603/PiAP.2014.0070. PMID 25339563
- [Background] Dowman L, McDonald CF, Hill CJ, Lee A, Barker K, Boote C, Glaspole I, Goh N, Southcott A, Burge A, Ndongo R, Martin A, Holland AE. Reliability of the hand held dynamometer in measuring muscle strength in people with interstitial lung disease. Physiotherapy. 2016 Sep;102(3):249-55. doi: 10.1016/j.physio.2015.10.002. Epub 2015 Oct 22. PMID 26596172
- [Background] Singer JP, Chen J, Blanc PD, Leard LE, Kukreja J, Chen H. A thematic analysis of quality of life in lung transplant: the existing evidence and implications for future directions. Am J Transplant. 2013 Apr;13(4):839-850. doi: 10.1111/ajt.12174. Epub 2013 Feb 22. PMID 23432992